CLINICAL TRIAL: NCT06948292
Title: Role of QRX-3 a Novel NAD Modulator in Ambulatory Chronic Kidney Patients
Brief Title: Role of QRX-3 in Chronic Kidney Disease Patients in Outpatients Clinics
Acronym: QRX-3 in CKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ebima Clifford Okundaye (Industry)
Responsible Party: Sponsor-Investigator, Ebima Clifford Okundaye, Principal investigator, Neukidney Inc.
Organization: Neukidney Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0002B
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease Stages 3-5; Diabetic Kidney Disease; Hypertensive Kidney Disease
Keywords: CKD; estimated GFR (eGFR); proteinuria; random urine protein creatinine ratio; creatinine change
MeSH Terms: conditions — Diabetic Nephropathies; Hypertensive Nephropathy; Proteinuria

STUDY DESIGN:
Intervention Model Description: QRX-3 added to intervention group in addition to standard therapy
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control group (No Intervention): control group - continued on standard therapy for CKD
- Intervention group (Active Comparator): QRX-3 drug given in addition to standard therapy for CKD
  Interventions: Drug: QRX-3

INTERVENTIONS:
Drug: QRX-3 — phase 2B CKD study
  Arms: Intervention group

SUMMARY:
QRX-3, a new drug that stabilized the kidney renal tubular cell and increase the activity of NAD ( nicotinamide adenine dineuclotide )within the kidney cells; leading to decrease oxidative changes intracellularly, repair of renal tubular injury and restoration of optimized renal function above baseline , will be studied in patients with progressive chronic kidney disease over 12 months . The result of the change in renal function expressed as creatinine GFR (Glomerular filtration decline) over the treatment duration will be compared in the treatment group will be compared to control group without the medication during that same period .

ELIGIBILITY:
Inclusion Criteria:

* Patient with Chronic kidney disease stage 3-5
* Estimated Glomerular function by MDRD of less than 60mls/min
* Patients with declining renal function ( as measured by eGFR by MDRD )
* Rate of decline of eGFR over the last one year of less than 20%
* Negative Serology markers for CKD etiology
* Provider perceived adherence to study follow- up

Exclusion Criteria:

* Rapid rate of decline in kidney function of > 10 % over 3 months
* Symptomatic renal failure
* Presence of any suspected Acute renal failure superimposed
* Presence of cast , hematuria, or abnormal urinalysis outside of simple UTI
* No known reversible cause of renal decline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
daily change in glomerular filtration rate by creatinine in mls/min | 12 months
  mean change in glomerular filtration rate by creatinine in mls/min in one year compare to baseline at screening

SECONDARY OUTCOMES:
change in proteinuria by mg/g | 12 months
  change in mean proteinuria measured by random urine protein/creatinine ratio at 12 months compare to control will be compared in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Neukidney Inc, Pasedena, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
if requested , deidentifiable data can be shared
Supporting Information: CSR
Time Frame: 4/21/2025 to 10/21/2025